CLINICAL TRIAL: NCT06675604
Title: Data Collection to Design and Validate LEOPARD Predictive Models of Delisting in Liver Transplant Candidates
Brief Title: LEOPARD Training and Validation Data Collection Study
Acronym: LEOPARD TVDCS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: European Society for Organ Transplantation (ESOT)-European Liver and Intestine Transplant Association (ELITA)ELITA (Unknown); University of Luxembourg (Other); Italian National Transplant Centre (CNT) (Unknown); La Fe University hospital Valencia (HULAFE) (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP240880
Record Dates: First submitted 2024-10-21; First posted 2024-11-05 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Decompensated Liver Cirrhosis; Primary Biliary Cholangitis; Primary Sclerosing Cholangitis; Hepato-cellular Carcinoma
Keywords: Liver transplantation; predictive models; data collection cohort; liver transplantation candidates
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Cholangitis, Sclerosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Subset 1: Decompensated cirrhosis as primary diagnosis, irrespective of liver disease etiology
- Subset 2: Other chronic end-stage liver diseases requiring LT, to be listed under a MELD-based allocation system (examples: primary biliary cholangitis, primary sclerosing cholangitis etc…)
- Subset 3: Hepato-cellular carcinoma as primary diagnosis, whatever the etiology of the underlying liver disease with or without underlying cirrhosis

SUMMARY:
Intro:

The present clinical research protocol is part of the LEOPARD European project (Grant n° 101080964 Horizon Europe) which aims to design and validate new predictive models of mortality among liver transplantation (LT) candidates. MELD based-liver graft allocation systems have become increasingly inaccurate over the last decade to predict mortality/dropout of liver transplantation (LT) candidates on the waitlist (WL). Wide disparities in mortality/dropout on the WL also exist across European countries, ranging from 5 to 30% according to transplantation indications and countries. In this setting, the European Commission- Horizon Europe funded-LEOPARD project intends to design new, 2nd generation, AI-machine learning-based predictive models of delisting in LT candidates, to better serve on time patients with the highest risk of dropout on the WL and to improve equity of access to LT across Europe.

Hypothesis/Objective:

The scientific justification of the LEOPARD TVDCS is therefore to collect a large set of data in liver transplantation candidates listed in Europe a) to design and b) to validate LEOPARD 2nd generation AI-based predictive models of mortality/dropout The primary objective is to develop new predictive models of mortality/drop out on the waitlist in patients with decompensated cirrhosis, or other end-stage chronic liver diseases, and in patients listed for Hepato-cellular carcinoma (HCC).

Method:

Longitudinal multicenter prospective health care data collection cohort study in 2 sets : Training/development set : Prospective health care data collection in 3,000 patients listed in 50 centres across 7 countries and Validation set: Prospective health care data collection in 1,500 subsequent patients listed in the same 50 centres.

ELIGIBILITY:
Inclusion Criteria:

* Adult [age 18;70] patients listed for:

  * decompensated cirrhosis as primary diagnosis, irrespective of liver disease etiology (subset 1) OR
  * other chronic end-stage liver diseases requiring LT, to be listed under a MELD-based allocation system (examples: primary biliary cholangitis, primary sclerosing cholangitis etc…) (subset 2) OR
  * HCC* as primary diagnosis, whatever the etiology of the underlying liver disease with or without underlying cirrhosis (subset 3). (HCC diagnosed on Barcelona/EASL criteria or histologically proven. HCC meeting or not Milan criteria, as per center practice.)
* Patients registered on national waiting lists under the MELD offering schemes, regardless of extra MELD points and MELD exceptions are affected or not.
* Patient (or trusted person, family member or close relation, if the patient is unable to be informed) who has been informed and did not express opposition to data collection

(*Of note, enrolment of patients with T1 tumors (1 single tumor < 2 cm diameter) not amenable to loco-regional therapies because of decompensation, and prioritized under the MELD system, will be allowed in Subset 1.)

Exclusion Criteria:

* Tumor vascular invasion (portal or hepatic veins) evidenced by imaging at pre transplantation work-up, including portal vein thrombosis stage 1
* Extra-hepatic metastasis of HCC, as assessed by sectional imaging, functional imaging (18 FDG PET CT/MRI) or histologically proven
* Patients who are under safeguard of justice or tutorship or curatorship
* Patient on AME (state medical aid)
* Participation to LEOPARD PVC 1 study of WP2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients listed for :
  * Decompensated cirrhosis as primary diagnosis, irrespective of liver disease etiology (subset 1)
  * Other chronic end-stage liver diseases requiring LT, to be listed under a MELD-based allocation system (examples: primary biliary cholangitis, primary sclerosing cholangitis etc…) (subset 2)
  * Hepato-cellular carcinoma as primary diagnosis, whatever the etiology of the underlying liver disease with or without underlying cirrhosis (subset 3)
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2029-02-04 (Estimated)

PRIMARY OUTCOMES:
Clinical primary endpoint considered as the event of interest to be predicted will be a composite of number of participants with mortality or drop out for being too sick on transplantation waiting list. | 3 months after listing in subsets 1 & 2 ; 12 months after listing in subset3
  * 3-month mortality/dropout for being too sick after listing in subsets 1 and 2
  * 12-month mortality/dropout for being too sick (tumor progression) after listing in subset 3

SECONDARY OUTCOMES:
Number of participants with 6- and 9-month pre LT mortality dropout for being too sick (all subsets) | 6 and 9 months after listing
  Mortality (all subsets)
Causes of death/drop-out for being too sick | From date of inclusion until date of death from any cause or date of drop-out for being too sick, whichever came first, assessed up to 12 months
  Causes of death/drop-out (all subsets)
Incidence of delisting for patient's decision or clinical improvement | From date of inclusion until date of delisting for patient's decision or clinical improvement, assessed up to 12 months
  delisting for patient's decision or clinical improvement
Time from listing to death/dropout | From date of listing until date of death from any cause or date of drop-out for being too sick, whichever came first, assessed up to 12 months
  Duration from listing to death/dropout (days)
Time to transplantation | From date of listing until date of transplantation, assessed up to 12 months
  Duration from listing to transplantation (days)
Number of participants with 6-month and 12 month post LT survival in subsets 1 to 3 | 6 months and 12 months after liver transplantation
  Survival in Training cohort subsets 1 to 3
Number of participants with 12-month HCC recurrence in subset 3 | 12 months after liver transplantation
  HCC recurrence in Training cohort subset 3
Number of participants with 6-month post-LT survival (all subsets) | 6 month after liver transplantation
  Survival in Validation cohort all subsets
6-month transplant benefit (all subsets) | 6 months after liver transplantation
  Relevant comorbidities (diabetes, hypertension, stroke, coronary disease, cancers, alcohol and tobacco consumption) in Validation cohort all subsets

CONTACTS AND LOCATIONS:
Locations (22):
- Universitätsklinik für Allgemeinchirurgie, Klinische Abteilung für Transplantation, Vienna, Austria
- Department of Gastroenterology and Hepatology Universitair Ziekenhuis Gent, Ghent, Belgium
- France (16):
  - CHU Jean Minjoz Besançon, Department of Hepatology, Besançon
  - CHU Trousseau Tours, Department of Hepatology, Chambray-lès-Tours
  - CHU Beaujon, Department of Hepatology, Clichy
  - Hospital Henri Mondor, Department of Hepatology, Créteil
  - CHU Dijon, Department of Hepatology, Dijon
  - CHRU Huriez Lille, Department of Hepatology, Lille
  - CHU Lyon Croix Rousse, Department of Hepatology, Lyon
  - CHU La Timone AP-HM, Department of Hepatology, Marseille
  - CHRU Montpellier Saint Eloi, Department of Hepatology, Montpellier
  - CHU L'Archet Nice, Department of Hepatology, Nice
  - CHU La Pitié Salpêtrière, Department of Hepatology, Paris
  - CHU Bordeaux Haut Levêque, Department of Hepatology, Pessac
  - CHU Pontchaillou Rennes, Department of Hepatology, Rennes
  - CHRU Strasbourg, Chirurgie Hepato-bilio-pancreatique et transplantation hepatique Department, Strasbourg
  - CHU Purpan Toulouse, Department of Hepatology, Toulouse
  - CHU Paul Brousse, Department of Hepatology, Villejuif
- Universitätsklinikum Schleswig - Holstein | UKSH · Transplantation Medicine, Kiel, Germany
- Italian National Transplant Center, Rome, Italy
- Center for Liver Tumors Leiden of the Leiden University Medical Center (LUMC), Leiden, Netherlands
- Servicio de HepatologíaHospital Universitario y Politécnico La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared. Datas are own by Assistance Publique-Hôpitaux de Paris (AP-HP), please contact sponsor for further information.